CLINICAL TRIAL: NCT05214131
Title: Randomized Study Of Novel Enuresis Alarm (GoGoband® )Vs Standard Nocturnal Enuresis Alarm (SNEA)
Brief Title: Randomized Study Of Novel Enuresis Alarm vs Standard Bedwetting Alarm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Southwest pediatric Device Consortium (Unknown); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000031281
Record Dates: First submitted 2022-01-25; First posted 2022-01-28 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Bedwetting; Nocturnal Enuresis; Urinary Incontinence
Keywords: bedwetting; biometric; artificial intelligence; machine learning; heart rate variability; nocturnal enuresis; enuresis; urinary incontinence
MeSH Terms: conditions — Nocturnal Enuresis; Urinary Incontinence; Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- gogoband alarm (Experimental): patients will be assigned to the novel bedwetting alarm
  Interventions: Device: gogoband
- standard nocturnal enuresis alarm (SNEA) group (Active Comparator): this is the standard bedwetting alarm that is presently available through out the world
  Interventions: Device: SNEA group

INTERVENTIONS:
Device: gogoband — use of biometric alarm to wake patient prior to wetting
  Arms: gogoband alarm
Device: SNEA group — standard bedwetting alarm is used to treat patients, alarm sounds after wetting accident has occurred
  Other Names: standard bedwetting alarm
  Arms: standard nocturnal enuresis alarm (SNEA) group

SUMMARY:
Identify the dry night rate in patients using the GoGoband® nocturnal enuresis device vs a standard Pflaundler bedwetting alarm.

DETAILED DESCRIPTION:
3.1 Problem Statement At the present time, there are no side-by-side comparison studies of GoGoband® vs SNEA. Since many of the prior studies were conducted using variable outcome parameters that makes direct comparisons of studies difficult it would be beneficial to obtain comparable data from the 2 groups and compare dry night rates for the 2 devices.

3.2 Purpose of Study/Potential Impact Our preliminary quality improvement data indicates that the GoGoband® is more efficacious than both medication and SNEA in an uncontrolled environment when deidentified data was analyzed off our servers. Our present database does not allow us to discern if patients are monosymptomatic nocturnal enuresis (MNE) or non monosymptomatic nocturnal enuresis (NMNE). Without this ability as well as for controlling for behavioral and academic problems which are known to affect outcomes in nocturnal enuresis studies, the investigators are not able to compare our results definitively and accurately to other treatment modalities.

Hypothesis Our hypothesis is that the GoGoband® is more effective than SNEA and Desmopressin in the treatment of Nocturnal Enuresis Primary Objective The primary objective of this study is to determine whether the GoGoband®] is as effective or more effective in comparison to children who use SNEA in a population of MNE patients with no underlying Attention deficit hyperactivity disorder (ADHD) in a 3 month period.

Secondary Objectives

To ascertain if familial incidence of nocturnal enuresis has an effect on outcomes

5.1 General Design Description The investigators propose the following study in patients who have been evaluated for primary nocturnal enuresis in our Yale New Haven Clinics.

* All patients to be evaluated for nocturnal enuresis will undergo standard evaluation and initial treatment for nocturnal enuresis which includes:
* Assessment Of Bowel Habits,
* Fill Out A Questionnaire To Evaluate For Voiding Dysfunction
* Treatment with routine bedwetting protocol of:

  1. Stopping drinks 1 HR before bedtime, meals at least 3 hrs before bedtime, eliminating milk and ice cream from dinner and on, making sure that bowel movements are occurring 4 times per week and treating appropriately if necessary.
  2. On return visit bedwetters and parents will be given the option of using medication , no further treatment, or alarm therapy.
  3. If patients choose alarm therapy, they will be asked if they wish to participate in the Randomized study comparing GoGoband® vs SNEA.
  4. Alarms will be provided to the patients free of cost to participants
  5. Patients in the alarm group will be treated for 3 months continuously.
  6. Patients in the SNEA group will record nightly if they wet their clothes and the report will be recorded and reviewed weekly
  7. GoGoband® patients' data will be automatically saved on the HIPPA Compliant servers and subsequently reviewed at the end of the week.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 6 to 21 years
4. In good general health as evidenced by medical history and diagnosed with MNE
5. Ability to and be willing to adhere to the treatment regimen. -

Exclusion Criteria:

1. No patient may have had treatment of MNE in the past 6 months whether with medications or alarms
2. Current use of on ADHD medications, Tricyclics, SSRI's, NRI's or any antipsychotic medications.
3. Presence of Autistic Spectrum disorder, ADHD, genetic syndrome associated with developmental or learning disabilities
4. Treatment with another investigational drug or other intervention within last 6 months
5. Any form of Diabetes Mellitus or Diabetes Insipidus
6. No patient with known Chronic renal disease with moderate to severe renal impairment (defined as a creatinine clearance below 50mL/min).
7. No patient with known hyponatremia or a history of hyponatremia.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Number of wet nights | 3 month period
  Comparison of alarms are to determine whether the GoGoband®] is as effective or more effective in comparison to children who use SNEA in a population of MNE patients with no underlying ADHD. The number of wet nights in each group will be compared to each other providing a comparison of the data. The gogoband group will be broken into two sections, training data and predictive and weaning data to compare against the SNEA data.
  Since the training data closely matches SNEA data, the investigators will compare the set of data and then compare the Predictive and Weaning data as the experimental group, since it has an active predictive alarm like the SNEA. The data will be compared using either a T test or Kruskal Wallis or anova depending on the number of comparisons performed and the data distribution is normal or not.

CONTACTS AND LOCATIONS:
Overall Officials: Israel Franco, MD, Principal Investigator — Dept of Urology, Yale School of Medicine
Locations (1):
- Yale New Haven Health, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website for the gogoband device — http://mygogoband.com